CLINICAL TRIAL: NCT00457873
Title: Isotonic Versus Hypotonic Saline for Maintenance Intravenous Fluid Therapy: A Pilot Randomized Trial
Brief Title: Isotonic Versus Hypotonic Fluid for Maintenance IV Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Bethany Foster, Principal investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PED-06-016
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Gastroenteritis; Bronchiolitis; Sepsis; Urinary Tract Infection
Keywords: surgery
MeSH Terms: conditions — Gastroenteritis; Bronchiolitis; Sepsis; Urinary Tract Infections | interventions — Sodium Chloride; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Experimental): 0.9% saline in 5% dextrose (intravenous)
  Interventions: Drug: 0.9% saline in 5% dextrose (intravenous)
- B (Active Comparator): 0.45% saline in 5% dextrose (intravenous)
  Interventions: Drug: 0.45% saline in 5% dextrose (intravenous)

INTERVENTIONS:
Drug: 0.9% saline in 5% dextrose (intravenous)
  Other Names: isotonic saline
  Arms: A
Drug: 0.45% saline in 5% dextrose (intravenous)
  Arms: B

SUMMARY:
Hyponatremia associated with administration of hypotonic intravenous (IV) fluids may have serious complications. It has recently been suggested that isotonic saline may be a more appropriate choice of maintenance IV fluid. This pilot and feasibility study aims to compare isotonic saline to 0.45% saline in hospitalized children requiring parenteral fluid support in order to:

Aim 1: To determine the feasibility of conducting a double-blind, randomized controlled trial comparing these solutions.

Aim 2a: To compare the rate of change in serum Na (mmol/L/hr) and the incidence of hyponatremia (Na <136 mmol/L) between patients receiving isotonic and hypotonic intravenous fluids at at least 50% of the traditional maintenance rate for an interval of at least 8 hours.

Aim 2b: To compare the incidence of adverse events between the two IV fluid treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* 1 month to 18 years of age
* Require IV fluids for at least 8 hr.
* Baseline serum sodium >=136 mmol/L & <=145 mmol/L

Exclusion Criteria:

* Baseline serum sodium concentration less than 136 mmol/L or greater than 145 mmol/L
* Renal disease, a history of cardiac dysfunction or evidence of cardiac dysfunction, pre-existing hypertension, diuretic use, edema, or known adrenal dysfunction
* Acute neurological illness such as meningitis or encephalitis
* Severe chronic neurological illnesses (uncontrolled seizure disorders, severe developmental delay)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
rate of change in serum sodium | 8 to 20 hours

SECONDARY OUTCOMES:
hypertension | 8 to 20 hours
congestive heart failure | 8 to 20 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bethany J Foster, MD, MSCE, Principal Investigator — Montreal Children's Hospital Research Institute
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Result] Hoorn EJ, Geary D, Robb M, Halperin ML, Bohn D. Acute hyponatremia related to intravenous fluid administration in hospitalized children: an observational study. Pediatrics. 2004 May;113(5):1279-84. doi: 10.1542/peds.113.5.1279. PMID 15121942
- [Result] Moritz ML, Ayus JC. Prevention of hospital-acquired hyponatremia: a case for using isotonic saline. Pediatrics. 2003 Feb;111(2):227-30. doi: 10.1542/peds.111.2.227. PMID 12563043
- [Result] Neville KA, Verge CF, Rosenberg AR, O'Meara MW, Walker JL. Isotonic is better than hypotonic saline for intravenous rehydration of children with gastroenteritis: a prospective randomised study. Arch Dis Child. 2006 Mar;91(3):226-32. doi: 10.1136/adc.2005.084103. Epub 2005 Dec 13. PMID 16352625
- [Derived] Saba TG, Fairbairn J, Houghton F, Laforte D, Foster BJ. A randomized controlled trial of isotonic versus hypotonic maintenance intravenous fluids in hospitalized children. BMC Pediatr. 2011 Sep 23;11:82. doi: 10.1186/1471-2431-11-82. PMID 21943218